CLINICAL TRIAL: NCT07061795
Title: The Effect of Home Visits on Healthy Lifestyle Behaviors During Pregnancy
Brief Title: Home Visits in Pregnancy and Healthy Lifestyle Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: serpil toker (Other)
Collaborators: Bilimsel Araştirma Projeleri Birimi, Tokat Gaziosmapaşa Üniversitesi (Unknown)
Responsible Party: Sponsor-Investigator, serpil toker, phd student, Tokat Gaziosmanpasa University
Organization: Tokat Gaziosmanpasa University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-KAEK-079
Record Dates: First submitted 2025-06-17; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Pregnancy; Prenatal Care; Home Visits
Keywords: Prenatal Care; Health Behavior; Maternal Health Services; Randomized Controlled Trial; Patient Education as Topic
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home visits group (Experimental)
  Interventions: Behavioral: healthy living behaviors
- routine follow-up (No Intervention): Healthy lifestyle behaviors of pregnant women given routine prenatal care

INTERVENTIONS:
Behavioral: healthy living behaviors — Effect of prenatal care with home visits on healthy lifestyle behaviors during pregnancy
  Arms: Home visits group

SUMMARY:
Abstract Background: Prenatal home visits allow early risk detection and comprehensive care in the pregnant woman's own environment.

Objective: To evaluate the effect of home-based prenatal care on health-promoting behaviors during pregnancy.

Design and Setting: A randomized controlled trial conducted at a family health center between September and December 2024.

Methods: A total of 200 pregnant women were randomly assigned to intervention (n=100) and control (n=100) groups. The intervention group received structured care via three monthly home visits; the control group received routine care. Data were collected using a personal information form and the Healthy Lifestyle Behaviors Scale in Pregnant (HLBS-P).

ELIGIBILITY:
Inclusion Criteria:

Gestational age less than 28 weeks Pregnancy record created by the Family Health Center

Exclusion Criteria:

Those who do not want to participate in the research Pregnant who do not speak Turkish

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — female gender
Enrollment: 200 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-28 (Actual)

PRIMARY OUTCOMES:
Health-promoting behavior score | Initially, second visit one month after baseline, third visit one month after second visit (There will be a total of 3 visits and it will last 3 months)
  The change in health-promoting behavior score measured by the ealthy Lifestyle Behaviors Scale in Pregnant Women (HLBS-P). This scale includes subdimensions such as pregnancy responsibility, hygiene, nutrition, physical activity, travel, and acceptance of pregnancy. The Cronbach's alpha reliability coefficients for the scale range between 0.79 and 0.94. Higher scores on the scale indicate healthier lifestyle behaviors among pregnant women.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpaşa Üniversitesi, Tokat Merkez, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared because the data include sensitive health information and participants did not consent to data sharing.